CLINICAL TRIAL: NCT06301126
Title: Effect of Virtual Reality on Pulmonary Function, Respiratory Muscle Strength and Functional Capacity After Upper Abdominal Surgeries
Brief Title: Virtual Reality on Pulmonary Function After Upper Abdominal Surgeries
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Morgan Allam, Assistant Professor of physical therapy for surgery, Faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004985
Record Dates: First submitted 2024-02-26; First posted 2024-03-08 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-05

CONDITIONS: Abdomen Hernia; Respiratory Complication
Keywords: Virtual reality; Pulmonary Function; Respiratory Muscle Strength; Functional Capacity; Upper abdominal surgery
MeSH Terms: conditions — Hernia, Abdominal

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual reality (Experimental): Participants will receive VR for 20 minutes followed by conventional physical therapy program for 45 minutes, 5 days/ week for 8 weeks.
  Interventions: Other: Virtual reality; Other: conventional physical therapy exercise program
- Control (Active Comparator): Participants will receive conventional physical therapy program (Deep diaphragmatic, costal breathing exercises, bronchial hygiene techniques and assisted cough) for 45 minutes, 5 days/ week for 8 weeks.
  Interventions: Other: conventional physical therapy exercise program

INTERVENTIONS:
Other: Virtual reality — The system included an Xbox 360® console, a sensor that detects motion (Kinect®), and a projector device with loudspeakers. The console, which was mounted on a table, reached 1 m tall. The Kinect® motion sensor was attached to the projector, which showed images onto a wall 2.5 metres distant from the playing field. The playing field was at least 1.8 m wide and 1.8 m long, with the Kinect® sensor situated 1.2 m away. The device was calibrated before each training session to accurately follow the motions of each subject.
  Arms: Virtual reality
Other: conventional physical therapy exercise program — Participants will receive conventional physical therapy exercise program (Deep diaphragmatic, costal breathing exercises, bronchial hygiene techniques and assisted cough) for 45 minutes, 5 days/ week for 8 weeks.

SUMMARY:
After upper abdomen surgery, respiratory muscle dysfunction is well recognised. After laparotomy and even laparoscopy, maximum static inspiratory and expiratory pressures are lowered, and recovery can take several days. A variety of reasons have been implicated in such respiratory muscle dysfunction, including irritation and inflammation, as well as injuries near the diaphragm, resulting in local mechanical failure, reflex inhibition, and pain.

DETAILED DESCRIPTION:
Virtual reality (VR) encourages an environment that attempts to create a moment of entertainment, motivation, and enjoyment with a variety of stimuli, with movements that stimulate physical and cognitive development, as well as the patient's active participation in the rehabilitation process. It is possible to assist in the alleviation of pain using the platform, at a low cost, through the playfulness given during rehabilitation, with an effective consumption of oxygen, range of motion, and use of the respiratory muscles more efficiently.

Participants with upper abdominal surgery will be randomly distributed into Group A (VR Group) which will receive VR for plus conventional physical therapy program and Group B (Control Group) which will receive conventional physical therapy program.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergone open upper abdominal surgery (hernia repair, cholecystectomy, large bowel removal, conventional laparotomy)
2. no prior surgical intervention for esophageal, gastric, or biliary tract resection
3. age 18-60 years
4. acceptable physical condition (permitting pulmonary function and functional capacity test).

Exclusion Criteria:

1. Cerebrovascular disease
2. use of immunosuppressants within 30 days of surgery
3. cardiovascular instability
4. chest physical therapy within the 8 weeks preceding study enrollment
5. visual impairment or hearing impairment;
6. bed-ridden patients;
7. any lung disorders
8. insulin-dependent diabetes mellitus
9. less than 6-months post thoracic or cardiac surgery
10. musculoskeletal impairment
11. cognitive disorders
12. Patients undergoing laparoscopic surgery as this induces smaller changes in the postoperative breathing mechanics than laparotomy does
13. heavy smokers or alcoholism

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Forced vital capacity (FVC) | 8 weeks
  FVC will be measured by using spirometer.

SECONDARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) | 8 weeks
  FEV1 will be measured by using spirometer.
Peak expiratory flow (PEF) | 8 weeks
  PEF will be measured by using spirometer.
Respiratory muscle strength | 8 weeks
  The inspiratory muscle strength will be verified by means of the maximum inspiratory pressure (MIP) and the expiratory muscular strength by means of maximum expiratory pressure (MEP) by using the digital Manovacuometer.
diaphragmatic mobility | 8 weeks
  Diaphragmatic mobility will be assessed using a high resolution ultrasound machine with a convex probe of 3.5 MHz on the right subcostal area in perpendicular incidence to craniocaudal axis in the assessment.
Functional capacity | 8 weeks
  Functional capacity will be measured by using 6-Minute Walk Test (6-MWT) that measures the maximum distance walked in a period of 6 min to assess the submaximal level of the functional capacity of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Hadaya M Eladl, PhD, Study Chair — Assistant professor of physical therapy for surgery, Faculty of physical therapy; Nabil M Abdel-Aal, PhD, Study Director — Assistant professor of physical therapy for basic sciences, Faculty of physical therapy
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study results
Supporting Information: Study Protocol, ICF
Time Frame: 6 months after publication
Access Criteria: Study protocol